CLINICAL TRIAL: NCT05193721
Title: A Clinical Study of the Safety and Tolerability of SHR-1901 in Subjects With Advanced Malignant Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1901-I-101
Record Dates: First submitted 2021-12-02; First posted 2022-01-18 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): SHR-1901 dose escalation at 0.1 mg/kg or 0.3 mg/kg or 1 mg/kg or 3 mg/kg or 10 mg/kg
  Interventions: Drug: SHR-1901

INTERVENTIONS:
Drug: SHR-1901 — SHR-1901 dose escalation at 0.1 mg/kg or 0.3 mg/kg or 1 mg/kg or 3 mg/kg or 10 mg/kg

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of SHR-1901 in subjects with advanced malignant tumors.To explore the reasonable dosage of SHR-1901.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced malignant tumors confirmed pathologically;
2. Failure of adequate standard treatment, or no effective standard treatment;
3. The expected survival period is more than 3 months;
4. The Eastern Cooperative Oncology Group (ECOG) physical fitness score is 0 - 1;
5. Have sufficient bone marrow and organ function (have not received blood transfusion or hematopoietic stimulating factor treatment within 14 days):(1)Neutrophil count (ANC) ≥ 1.5×10e9/L; (2)Platelet count (PLT) ≥90×10e9/L; (3)Hemoglobin (Hb) ≥ 9.0g/dL; (4)Serum creatinine ≤1.5 times the upper limit of normal (ULN) or creatinine clearance ≥60 ml/min (calculated using Cockcroft-Gault formula); (5)Total bilirubin (BIL) ≤1.5 times the upper limit of normal (ULN), patients with liver cancer/liver metastasis should be ≤2×ULN; (6)Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) levels ≤ 3 times the upper limit of normal (ULN), patients with liver cancer/liver metastasis ≤ 5×ULN; (7)International normalized ratio (INR) ≤ 1.5, prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤ 1.5 times ULN;
6. Female subjects of childbearing age must undergo a serum pregnancy test within 3 days before starting the study medication, and the result is negative, and are willing to use a medically approved high-efficiency contraception during the study period and within 6 months after the last administration of the study drug Measures: For male subjects whose partners are females of childbearing age, they should be surgically sterilized, or agree to use effective methods of contraception during the study period and within 3 months after the last study administration;
7. With my consent and signed informed consent form, I am willing and able to comply with planned visits, research treatments, laboratory inspections and other test procedures.

Exclusion Criteria:

1. Subjects have clinically significant cardiovascular/cerebrovascular diseases, such as: cerebrovascular accident/stroke within 6 months before entering the study, myocardial infarction within 6 months before entering the study, unstable angina pectoris, NYHA level 2 or higher Patients with heart failure and clinically significant supraventricular or ventricular arrhythmia in need of treatment or intervention;
2. The subject has any active autoimmune disease or a history of autoimmune disease (such as the following, but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, nephritis, vasculitis, decreased thyroid function [ Subjects who do not require medication or can be controlled by hormone replacement therapy only can be included]; subjects who have vitiligo or asthma has been completely relieved in childhood, and those who do not need any intervention after adults can be included; subjects who need bronchiectasis Asthma for medical intervention cannot be included);
3. Known to be allergic to the study drug or any of its excipients, or have a severe allergic reaction to other monoclonal antibodies;
4. He had other active malignant tumors within 2 years before entering the study. Except for skin basal cell or squamous cell carcinoma, superficial bladder cancer, cervical carcinoma in situ, intraductal carcinoma in situ of the breast, and papillary thyroid carcinoma that can be treated locally and have been cured;
5. There is a large amount of fluid in the serous cavity that requires repeated puncture or drainage;
6. There are major acute or chronic infections, including:
7. Active bacterial or fungal infections requiring systemic treatment;
8. Active tuberculosis (tuberculosis, TB) or subjects with a history of active tuberculosis infection ≤48 weeks before screening, regardless of treatment;
9. Human immunodeficiency virus (HIV) infection or known acquired immunodeficiency syndrome (AIDS);
10. Untreated active hepatitis (hepatitis B, defined as HBV-DNA ≥ 2000 IU/ml or ≥ 104 copy/ml; hepatitis C, defined as HCV-RNA higher than the detection limit of the analysis method) or combined with hepatitis B and Co-infection of hepatitis C;
11. During the screening period/before the first administration, fever of unknown origin> 38.5°C (according to the judgment of the investigator, fever caused by tumor can be included in the group);
12. Participated in or are participating in other clinical studies within 4 weeks before starting the study drug treatment (subjects who have entered the follow-up period are calculated based on the time of the last use of the experimental drug or device);
13. Has a history of psychotropic drug abuse or drug abuse. There are other serious physical or mental illnesses or laboratory abnormalities that may increase the risk of participating in the research, or interfere with the results of the research, as well as patients who the researcher believes are not suitable for participating in this research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety endpoints: Number of subjects with adverse events and the severity of adverse events | every 4 weeks after treatment initiation（through study completion，average 5 months)
DLT | during the first 28-day cycle of SHR-1901 treatment
MTD | 4 weeks after treatment initiation
RP2D | 4 weeks after treatment initiation

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided